CLINICAL TRIAL: NCT06407401
Title: Improvement of Quality of Life Through Supportive Treatments for Hormone Therapy - Related Symptoms in Patients With Early Breast Cancer; A Pragmatic Randomized Controlled Trial
Brief Title: Improvement of Quality of Life Through Supportive Treatments for Hormone Therapy - Related Symptoms in Patients With Early Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EORTC-2237-BCG-QLG
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: ER+ Breast Cancer; HER2-negative Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Drug-Related Side Effects and Adverse Reactions; Musculoskeletal Pain
Keywords: Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions; Musculoskeletal Pain | interventions — Duloxetine Hydrochloride; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (SoC) (Active Comparator): Standard of care (SoC) including a booklet focused on healthy behaviors
  Interventions: Behavioral: Booklet for healthy behaviors
- Experimental arm SoC with duloxetine (Experimental): Duloxetine 60 mg (1 pill a day) + SoC
  Interventions: Drug: Duloxetine 60 MG; Behavioral: Booklet for healthy behaviors
- Experimental arm SoC with Furosemide (Experimental): Furosemide 40 mg (1 pill a day) + SoC
  Interventions: Drug: Furosemide 40 mg; Behavioral: Booklet for healthy behaviors

INTERVENTIONS:
Drug: Duloxetine 60 MG — Patients randomized to the duloxetine arm will take duloxetine orally daily, with or without food, on a continuous dosing schedule.
  Initial dose is 30 mg daily for 1 week, followed by 60 mg daily for a total of 6 months of treatment, followed by a taper off the medication of 30 mg daily for 1 additional week.
  Arms: Experimental arm SoC with duloxetine
Drug: Furosemide 40 mg — Patients randomized to the furosemide arm will take furosemide 40 mg orally daily, on an empty stomach with plenty of liquid, on a continuous dosing schedule.
  Arms: Experimental arm SoC with Furosemide
Behavioral: Booklet for healthy behaviors — All patients will receive usual care, including a booklet focused on healthy behaviors, particularly physical exercise, to manage endocrine therapy side-effects.

SUMMARY:
This study is a pragmatic international, multicenter, randomized, open label 3- arm trial of standard care vs. two pharmacological interventions: duloxetine or furosemide in patients with stage I-III ER+/HER2- early breast cancer with joint, muscle and/or bone pain caused by the endocrine therapy.

The purpose of the BC-QOL trial is to find out whether treatment with duloxetine or furosemide, given while patients are on treatment with endocrine therapy, is active in improving quality of life (QoL), specifically by improving joint, muscle and/or bone pain caused by the endocrine therapy (based on EORTC QLQ-BR42 skeletal scale).

DETAILED DESCRIPTION:
Patients, identified by their clinicians as suffering from Grade 2 or above endocrine therapy-related musculoskeletal symptoms [joint/bone/muscle pain]) for, at least, 4 weeks before enrolment will be centrally randomized 1:1:1 between:

* Control arm: Standard of care (SoC) including a booklet focused on healthy behaviors
* Experimental arm: Duloxetine 60 mg (1 pill a day) + SoC
* Experimental arm: Furosemide 40 mg (1 pill a day) + SoC

Treatment duration will be 6 months. All patients will receive usual care, including a booklet focused on healthy behaviors, particularly physical exercise, to manage endocrine therapy side-effects. Treatment administration and modifications as well as specific monitoring should be done in accordance to the SmPC of the corresponding drugs.

ELIGIBILITY:
Inclusion criteria:

* Female (both pre- and postmenopausal) or male patients
* Age ≥18 years
* Ongoing adjuvant ET (tamoxifen or OFS plus tamoxifen or OFS plus AI or AI ) for ER positive HER2 negative breast cancer stages I-III
* Patients must have received at least 3 months and up to 3 years of ET and planned to continue ET during the study conduction
* Present endocrine therapy related MSK pain (arthralgia and/or bone pain and/or myalgias), evaluated by the treating clinician as at least grade 2 CTCAE V5.0 for, at least, 4 weeks before enrolment, at the time of the clinic visit:

  * Grade 2: moderate pain; limiting instrumental activities daily living (ADL)
  * Grade 3: severe pain; limiting activities self-care ADL
* Previous chemotherapy is allowed if completed at least 3 months before enrolment
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Adequate organ function
* Completed baseline assessment of patient-reported questionnaires (EORTC QLQ-C30 and EORTC QLQ breast module)
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to the first dose of study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, except for those who had prior hysterectomy). However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression, or other reasons.

* Patients of childbearing / reproductive potential must agree to use at least one acceptable effective contraceptive measure until treatment discontinuation.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 1 month after the last study treatment.

Exclusion criteria:

* Current history of moderate/severe depression and/or anxiety, both defined as grade≥2 CTCAE V5.0
* History of suicide-related events
* Current use of diuretics, antidepressants and/or phytoestrogens
* Current use of prescribed or natural medicines with known interactions with furosemide and/or duloxetine
* Contraindications to duloxetine:

  * Severe renal impairment (creatinine clearance < 30 mL/min)
  * Uncontrolled hypertension
  * Hepatic impairment Child Pugh Class B or C
* Contraindications to furosemide:

  * Symptomatic hypotension, hypovolemia, or dehydration
  * Severe renal impairment (creatinine clearance < 30 mL/min)
  * Severe hypokalaemia and/or severe hyponatremia
  * Addison's disease
  * Porphyria
* Uncontrolled intercurrent illness, including psychiatric conditions, chronic alcoholism, and drug addiction, that would, in the judgment of the investigator, limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Known difficulty in tolerating oral medications or conditions which would impair absorption of oral medications such as: uncontrolled nausea or vomiting (i.e., CTCAE ≥ Grade 3 despite antiemetic therapy), ongoing gastrointestinal obstruction/motility disorder, malabsorption syndrome, or prior gastric bypass
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol, understanding and completion of questionnaires and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the trial.
* Participation in another interventional study with drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-04-18 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Endocrine therapy related musculoskeletal pain | 3 months
  Assessed by the Skeletal scale from the EORTC-QLQ-BR42 questionnaire, with the minimum and maximum values being 0 - 100 and higher score means worse outcome.

SECONDARY OUTCOMES:
Endocrine therapy related musculoskeletal pain | 6 months
  Assessed by the Skeletal scale from the EORTC-QLQ-BR42 questionnaire, with the minimum and maximum values being 0 - 100 and higher score means worse outcome.
Overall quality of life | 3 months and 6 months
  Assessed by the Global Health status/Quality of Life scale from the EORTC-QLQ-C30 questionnaire, with the minimum and maximum values being 0 - 100 and higher score means better outcome.
Emotional functioning | 3 months and 6 months
  Assessed by the emotional functioning scale from the EORTC-QLQ-C30 questionnaire, with the minimum and maximum values being 0 - 100 and higher score means better outcome.
Endocrine therapy related symptoms | 3 months and 6 months
  Assessed by the endocrine therapy symptom scale from the EORTC-QLQ-BR42 questionnaire, with the minimum and maximum values being 0 - 100 and higher score means worse outcome.
Discontinuation of endocrine therapy | 6 months
  Proportion of patients who discontinued endocrine therapy